CLINICAL TRIAL: NCT04379856
Title: A Phase I/II Proof of Concept, Open-Label, Repeat Dose, Dose Escalation Study of NM-002 in Adult Patients With Short Bowel Syndrome (SBS)
Brief Title: Proof of Concept Study in Patients With Short Bowel Syndrome
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: 9 Meters Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NMSBS01-001
Record Dates: First submitted 2020-04-02; First posted 2020-05-08 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose 1 (Experimental): NM-002 will be administered at the indicated dose by subcutaneous injection on Days 1 and 15.
  Interventions: Drug: NM-002
- Dose 2 (Experimental): NM-002 will be administered at the indicated dose by subcutaneous injection on Days 1 and 15.
  Interventions: Drug: NM-002
- Dose 3 (Experimental): NM-002 will be administered at the indicated dose by subcutaneous injection on Days 1 and 15.
  Interventions: Drug: NM-002

INTERVENTIONS:
Drug: NM-002 — NM-002 is a fusion protein, of which the pharmacological active portion is the glucagon-like peptide-1 (GLP-1) analog domain with the same amino acid sequence as the active pharmaceutical ingredient (exenatide)

SUMMARY:
This is a Phase I/II. proof of concept, open label, two-dose, dose escalation study of NM-002 in adult patients with SBS who previously responded to exenatide. NM-002 is planned to be administered twice, at up to 3 different dose levels, in up to 3 cohorts, each consisting of 3-4 patients. Doses will be administered on Days 1 and 15 by subcutaneous injection. Patients will be monitored for their usage of parenteral supplementation, and will fill out a daily diary for their symptoms of SBS. Urine output will be measured on a daily basis. Patients will be followed for 6 weeks after the second dose.

DETAILED DESCRIPTION:
During a baseline period, all subjects will remain on their current prescription for administration of PS. Between Days -7 to -5 patients who have met initial screening criteria will return to the clinic and be enrolled into the study. Patients will be trained on diary usage and patients receiving the SBS meds will be instructed to discontinue use of their medications; Imodium, lomotil, and opium tincture.

On Day -4, subjects will begin diary entries. For 48 hours, on Days -1 and 0, patients will record in their diaries total urine output, PS usage, stool output and oral liquid intake.

On Study Day -1, patients will visit the clinic for baseline safety assessment, and review of symptoms of malabsorption and PS usage. Baseline SF36 and Bowel Symptom questionnaires will be administered.

On Day 1 of treatment, patients will return to the clinic with a sample of urine collected during the baseline run-in for urinalysis. They will have blood samples drawn for clinical laboratory assessment and for pre-dose PK levels, anti-drug antibody, and AE assessments. Following administration of study drug on Day 1, subjects will undergo additional serial PK blood draws.

Serial blood samples for the pharmacokinetic evaluation of NM-002 will be drawn on Days 1 and 15, with single samples obtained on 2, 3, 4, 5, 8, 16, 17, 18, 19, 22 and 29. Additional blood samples will be taken for clinical laboratory evaluations.

Blood glucose meters will be provided to patients to record their daily blood glucose levels, and to check their blood glucose should any symptoms related to hypoglycemia occur. Patients will receive written instructions regarding the symptoms of hypoglycemia and how to manage them at home. They will be provided with glucose gel tubes and instructed in their use.

At any time on Days 6 through 24, the investigator may call for a reduction or increase in PS, based on patient diary data and his/her clinical judgment. If a change in PS occurs, serum electrolytes will be assessed within 48 hours of implementing the change in PS.

If patients have experienced a reduction in PS administration during the study, on Day 25 they will be returned to their pre-study, standard PS regimen. On Day 27, patients will be asked to return to their individual oral liquid intake established during the baseline run-in period, and they will record their urine output volume for 48 hours (on Days 27 and 28).

Any patients who experience an increase in PS administration over the original baseline level will remain on the new level of PS on Days 27 and 28.

Patients will return to the clinic on Day 29. Blood samples will be drawn for clinical laboratory analysis and for PK. Patients will continue to make daily diary entries through Day 55. Telephone follow-ups will be conducted by the investigational site on Days 35±1 and 42±1 to assess any requirement for PS adjustment.

Patients will return to the clinic on Day 56 ± 2 for a final safety assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females with SBS secondary to surgical resection of small intestine, with or without an intact colon
2. 18-75 years of age at the time of screening
3. Female subjects must be postmenopausal (at least 2 years prior to dosing) or surgically sterile or agree to use an acceptable form of birth control from screening until 30 days after last dose. If oral contraceptives are used, Subject must have been on a stable dose for ≥6 months. (See below, "Participation of Women", for additional detail.)
4. Male subjects must agree to use an acceptable form of birth control during the study and for 90 days after the last dose. Male subjects may not donate sperm for 90 days after last dose.
5. At least 6 months since last surgical bowel resection
6. Patients may be on Parenteral support (nutrition and/or fluid and electrolytes [PS]) for at least some of their nutritional needs.
7. If on PS, stable administration of PS volume for 1 month (±20% vol) prior to enrollment.
8. Able to ingest solid foods and drink
9. Willing to adhere to a defined oral intake of fluids on certain days as required by protocol and based on the individual's routine daily consumption.

Exclusion Criteria:

1. Positive results on the HIV, Hepatitis, or drug screens.
2. Pregnancy or lactation
3. Body mass index <18 or >30 kg/m2
4. Clinically significant intestinal adhesions and/or chronic abdominal pain
5. Active Crohn's disease or IBD (as evaluated by standard procedures employed by the investigator/institution). If in remission, must be ≥12 weeks of remission prior to enrollment.
6. If on chronic systemic narcotics, the patient must have been on a stable dose for >12 weeks
7. Inflammatory bowel disease patients who have NOT been on a stable drug treatment regimen for at least the past 3 months.
8. Visible blood in the stool within the last 3 months
9. Catheter sepsis experienced within the last 3 months
10. Known heart failure or active coronary disease
11. Known celiac disease
12. Radiation enteritis, scleroderma, coeliac disease, refractory or tropical sprue, diabetes
13. Alcohol or drug abuse within the last 12 months
14. Inadequate hepatic function as defined by: ALT and ASAST both >2.0X ULN; TBL >2X ULN; or ALP >2.5X ULN
15. Inadequate renal function as defined by serum creatinine <0.7 or >1.3 mg/dL (in men) and <0.6 or >1.1 mg/dL in women.
16. Personal or family history of medullary thyroid cancer.
17. History of pancreatitis.
18. Any patient who receives insulin in their PS.
19. Any hospitalization within 1 month before screening visit
20. Systemic corticosteroids, methotrexate, cyclosporine, tacrolimus, sirolimus, infliximab, or mycophenolate mofetil (CellCept®) within 30 days of screening
21. Any use of growth hormone, or growth factors such as native GLP-2 or GLP-2 analog (teduglutide) within the last 3 months
22. Use of antibiotics within the last 30 days
23. Subject not capable of understanding or not willing to adhere to the study visit schedules and other protocol requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-06-23 (Actual); Primary Completion 2020-12-11 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of repeated doses of NM002 three different dose levels | 56 days
  Assess adverse event profile of each dose and dose level

CONTACTS AND LOCATIONS:
Locations (1):
- Research Facility One, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No